CLINICAL TRIAL: NCT05108025
Title: A Study Of The Tolerability, Safety, And Efficacy Of DMT310 For The Treatment Of Acne Rosacea
Brief Title: DMT310-005 Topical in the Treatment of Acne Rosacea
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dermata Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMT310-005
Record Dates: First submitted 2021-10-26; First posted 2021-11-04 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Acne Rosacea
MeSH Terms: conditions — Rosacea | interventions — Powders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Treatment 1 (Experimental): DMT310 Powder mixed with Hydrogen Peroxide
  Interventions: Drug: Topical Powder
- Study Treatment 2 (Experimental): Placebo powder mixed with Hydrogen Peroxide
  Interventions: Drug: Placebo Topical Powder

INTERVENTIONS:
Drug: Topical Powder — Topical Powder mixed with diluent
  Arms: Study Treatment 1
Drug: Placebo Topical Powder — Placebo Topical Powder mixed with diluent
  Arms: Study Treatment 2

SUMMARY:
The objective is to evaluate the tolerability, safety, and efficacy of DMT310 topical powder mixed with diluent in male and female patients with moderate to severe facial acne rosacea.

ELIGIBILITY:
Inclusion Criteria:

Patient is male or non-pregnant female at least 18 years of age.

Clinical diagnosis of moderate to severe papulopustular acne rosacea as determined by:

Investigator's Global Assessment (IGA) at Randomization score of 3 or 4. Patient has at least 15 inflammatory lesions on the face

Patient is willing to apply the Investigational Product as directed

Patient is willing and able to comply with the protocol

Exclusion Criteria:

Patient is pregnant or planning to become pregnant Patient is taking a topical therapy on the face which may affect the patient's rosacea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy as measured by lesion counts | 12 Weeks
  Inflammatory lesion counts
Efficacy as measured by Investigator Global Assessment (IGA) | 12 Weeks
  IGA Scale:
  0 Clear No papules and/or pustules
  1. Almost Clear Rare papules and/or pustules
  2. Mild Few papules and/or pustules
  3. Moderate Pronounced number of papules and/or pustules (but less than numerous papules and/or pustules)
  4. Severe Numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | 12 Weeks
  Incidence of adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Dermata Investigational Site, Austin, Texas, United States